CLINICAL TRIAL: NCT06935825
Title: Respiratory Muscles in End-stage Lung Disease: PAthophysiological Processes & Clinical Consequences
Acronym: Re-MAP
Status: Not yet recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Erasmus Medical Center (Other); Amsterdam UMC, location VUmc (Other); Radboud University Medical Center (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: PaNaMaID: 22059
Record Dates: First submitted 2025-04-03; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: COPD
Keywords: COPD; NIV; Lung transplantation; Respiratory muscles; diaphragm; ultrasound; sEMG; MIP
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — To study the respiratory myofibers, we will obtain muscle biopsies of diaphragm and intercostal muscles during LTx. From the biopsies individual myofibers will be isolated and their structure and contractility will be assessed. After the isolation of individual myofibers, the remaining muscle tissue will be used for immunohistochemical staining and gene expression analyses to study the molecular mechanisms underlying respiratory muscle dysfunction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- NIV+: Group of patients on nocturnal NIV prior to LTx
- NIV-/hypercapnic: Group of patients who are chronic hypercapnic but not on NIV prior to LTx
- normocapnic: Group of normocapnic patients prior to LTx

SUMMARY:
Rationale: In patients with chronic lung diseases, the role of respiratory muscle dysfunction has been underestimated. Also, current treatment options, like chronic NIV and lung transplantation (LTx), might also have deleterious effects on the respiratory muscles, and the mechanisms are poorly understood.

Therefore in this exploratory study the objectives are to:

1. Determine in vivo respiratory muscle function and progression of respiratory muscle dys-function in end-stage COPD patients
2. Establish the correlation between changes in the structure and contractility of respiratory myofibers and in vivo respiratory muscle function.
3. Establish the effect of chronic NIV on structure and contractility of respiratory muscle fi-bers
4. Determine whether the structure and contractility of respiratory muscles cells at the time of LTx predicts clinical recovery post-LTx.

Study design: The study will be an exploratory observational cohort study following patients on the LTx waiting list during the waiting period and afterwards until they showed functional recovery of respiratory muscle function.

Study population: Adult COPD patients on the LTx waiting list will be included. Intervention (if applicable): None

Main study parameters/endpoints:

To assess clinical functioning of the respiratory muscles we will assess respiratory electrical activity as a measure of respiratory effort by surface EMG, and thickening fraction of the diaphragm and intercostal muscles and diaphragm excursions by ultrasound and maximal in- and expiratory pressure to assess muscle output; all before and after LTx. We will relate and correct these data for hyperinflation and degree of lung damage by using data from standard care lung function tests and CT scans, and will relate these measurements to prior treatment (NIV settings) and outcome after LTx, by retrieving these data from the EPD.

To assess contractility of respiratory myofibers and in vivo respiratory muscle function, biopsies will be taken during LTx surgery and the biopsies will be analyzed in the lab of Prof. Ottenheijm (AmsterdamUMC) for individual myofiber functioning (strength, calcium sensitivity, myofiber characteristics) and in the lab of Dr. Pouwels for extracellular matrix characteristics.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Overall, risks are believed to be minimal. The clinical measurements are non-invasive and/or regular performed in clinical practice. Also, we decided to do those measurements during regular control visits, limiting the burden for the patients. Taking biopsies from the respiratory muscles during surgery has been extensively performed without any risk; the biobank of the Ottenheijm group contains > 500 samples and never any complication has been observed. Also, in preparation of the present study we performed a pilot study in 12 COPD patients of whom.. biopsies were taken at the UMCG without side effects or complications. The biopsies will be done with the patients being under full anesthesia, so participants will feel no discomfort.

DETAILED DESCRIPTION:
Considering that a) there is a substantial proportion of patients with severe COPD that develop respiratory muscle dysfunction-induced CHRF; b) respiratory pump failure results in significant morbidity and mortality; and c) the response to current treatment options is highly variable, presumably due to detrimental effects on the respiratory muscle pump, there is a high need for research identifying the pathophysiological mechanisms that underlie respiratory muscle dysfunction in end stage COPD. To meet this need, we will combine in vivo respiratory muscle testing with studies on unique respiratory muscle biopsies to test the hypothesis that respiratory muscle dysfunction is caused by atrophy and reduced contractility of single respiratory myofibers, and that this underlies the development of CHRF. Furthermore, we will test the hypothesis that respiratory muscle dysfunction is exacerbated by NIV and contributes to difficulties in post-LTx recovery. The outcomes will identify targets for intervention and prevention of CHRF.

ELIGIBILITY:
In order to be eligible to participate in this study, a participant must meet all of the following criteria:

* Age > 18 years old
* Severe COPD defined as COPD GOLD stage III or IV (FEV1 < 50% of predicted; FEV1/FVC ratio < 70%, no significant reversibility, smoking history of at least 10 pack-years).
* Being on the lung transplant waiting list
* Being able to understand the patient information and provide written informed consent for participation in the study

A potential participant who meets any of the following criteria will be excluded from participation in this study:

* Patients suffering from acute conditions at the time of inclusion or LTx
* Patients using more than 20 mg of morphine, or an equivalent, or more than 20 mg oxazepam, or an equivalent, at the time of inclusion or LTx

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: COPD patients on the lung transplantation waiting list
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory neural drive | 3-6 monthly before LTx, directly before and after LTx, 3-6 monthly after LTx
  With surface EMg (sEMG) a measure of respiratory neural drive is obtained, which could be used as stand alone parameter to estimate effort and, when combined with output parameters as diaphragm movement or MIP/MEP, might be useful to estimate neuro-ventilatory efficiency.
Respriatory muscle output - contraction and movement | 3-6 monthly before LTx, directly before and after LTx, 3-6 monthly after LTx
  With ultrasound, we will measure diaphragm and intercostal thickening fraction (DF-TF) thereby investigating the amount of muscle contraction. Diaphragm excursion will be measured from subcostally.
Respriatory muscle output - strength | 3-6 monthly before LTx, directly before and after LTx, 3-6 monthly after LTx
  Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) will be measured at the lung function department according to ERS guidelines or by using a handheld device when patients are at the ward. Patients are asked to inhale and exhale deeply against a resistance and then measuring airway pressure produced.
Myofiber mechanics | Biopsies are obtained during LTx
  The maximum force generating capacity, the force response to a range of submaximal [Ca2+], active stiffness (reflecting the number of attached and non-attached myosin heads) is determined of individual myofibers.
Low angle X-ray diffraction | Biopsies are obtained during LTx
  Measure the position of myosin heads in relaxed and in activated myofibers
Mant-ATP chase experiments | Biopsies are obtained during LTx
  To biochemically assess the percentage of myosin heads in the SRX state
Myofiber and extra-cellular matrix structure | Biopsies are obtained during LTx
  We will assess myofiber size by immunohistochemistry using antibodies that label the sarcolemma and myosin heavy chain isoforms
Transcriptomic and proteomic analyses of muscle biopsies | Biopsies are obtained during LTx
  To study the activation of fibrosis pathways we will apply RNAseq and proteomics on the biopsies

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Amsterdam University Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen
  - Radboud University Medical Center, Nijmegen
  - Erasmus Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: No
With such a specific group it is too difficult to keep it anonomyzed